CLINICAL TRIAL: NCT00308386
Title: Impact of Nurse Case Management on Diabetes Co-morbidities
Brief Title: DYNAMIC Study: (Diabetes Nurse Case Management And Motivational Interviewing for Change)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R18 67495 (completed); R18DK067495 (NIH)
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus; Hypertension; Hyperlipidemia
Keywords: Nurse Case Management; Diabetes; Hypertension; Hyperlipidemia; Behavior therapy; Motivational interviewing
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Nurse Case Management intervention — Intervention is meeting with nurse case managers

SUMMARY:
Although strong clinical evidence exists that patients with diabetes should achieve certain clinical goals (i.e. HbA1C, BP, LDL, etc.), to reduce morbidity and mortality national surveys indicate that only a minority of people with diabetes achieves these goals.

Hypothesis: combination of nurse case management and enhanced behavior change counseling will improve outcomes for glycemic control, blood pressure and cholesterol in high risk patients with Type 2 diabetes when compared to usual care over a 3 year period.

Study design- The study will be a three year randomized control trial that will select patients that have either A1C >8.5, LDL >130, or BP >140/90. Nurse case managers, trained in clinical guidelines and brief behavior change counseling techniques (motivational interviewing), will aim to foster patient adherence in the experimental group patients. Nurse case managers will use standing orders to set an implementation of clinical guidelines (for diabetes, hypertension, hyperlipidemia and depression) with individual follow up.

A total of 820 patients between the all 9 (6 Hershey Medical Center and 3 Reading Hospital affiliated clinics) will be sought. One third of the study patients will be recruited from the underserved Hispanic population in the Reading area. Patients will be randomized by physician i.e. one physician will be randomly assigned to have all their patients co-managed by a nurse case manager; the other will have usual care without any contact with nurse case manager.

Nurses will be trained and then initiate a small pilot study in July thru August. Full recruitment and initiation of study will begin in September 2006.

Clinic Activities - Each nurse will be responsible for 3 clinics. Nurses will work under the supervision of the primary care physicians. A set of clinical guidelines will be developed with physician input that will serve as the over-riding framework for the nurses.

Outcomes - Over a three-year period the investigators will evaluate clinical response (improvements in A1C, BP, LDL, and depression when present) as well as a series of other measures that will be obtained by surveys (patient satisfaction, quality of life, self-management behaviors). Provider satisfaction will be measured using a standardized tool. Finally, cost effectiveness of the intervention and evaluation of the potential barriers to implementation will be studied.

DETAILED DESCRIPTION:
1. Rationale: Diabetes mellitus is a prevalent disease and results in high health care expenditures, the majority of which are due to preventable complications of diabetes. Current evidence indicates that care of patients with diabetes mellitus falls short of the standards set by the American Diabetes Association and a large proportion of these patients do not achieve their treatment goals. Multiple ways to deliver care to patients with diabetes have been studies. The investigators propose a 3 year randomized-controlled study to assess impact of the combination of nurse case management (NCM) combined with enhanced behavior change counseling on glycemic control and co-morbidity outcomes in high-risk patients with Type 2 diabetes when compared to usual care
2. Key Objectives:

   Specific Aim 1. Determine the efficacy of an enhanced nurse case management (NCM) intervention to promote patient adherence leading to positive clinical outcomes (HbA1C, LDL, blood pressure, and process measures) in high-risk patients in primary care over a period of three years. High-risk patients with Type 2 diabetes will be recruited from 9 primary care clinics and randomized to NCM intervention vs. usual care. A major focus of this proposal is to test the efficacy of NCM in a minority population with high risk of poor outcomes (approximately 38 % of the study population will be Hispanic). The investigators anticipate a significant increase in percentage of patients reaching the goals for HbA1C (< 7.0%), BP (<130/80), LDL (<100 mg/dl) in patients in the NCM group compared to the control group of usual care. The investigators also hypothesize that there will be significant improvement in process measures (% patients having a yearly dilated eye exam, foot exam, urinary screen for microalbuminuria, aspirin use, lipid evaluation) and depression scores in patients in the NCM group compared to the control group of usual care.

   Specific Aim 2. Quantify the impact of enhanced nurse case management on health-related quality of life, patient satisfaction, self-management behaviors, and provider satisfaction. A unique feature of our study is to address the impact of our intervention on these critical outcomes, which have not been addressed in the existing NCM literature. The investigators anticipate improved adherence, lower levels of diabetes specific emotional distress, higher levels of diabetes specific quality of life, increased patient satisfaction with treatment, and improved provider satisfaction in the NCM group compared to the usual care group. The following surveys will be completed and analysed:the PAID survey looking at Emotional distress associated with diabetes, the ADDQOL (Diabetes specific quality of life) survey, the DTSQ (Patient satisfaction) survey and the SDSCA (Diabetes self care activities) survey.

   Specific Aim 3. Evaluate the cost-effectiveness of an enriched NCM intervention. The investigators expect that the NCM intervention will be effective in improving clinical outcomes for patients with type 2 diabetes; however, there may still be barriers to more widespread adoption unless the benefits of investing in or reimbursing for NCM can be justified by the costs. Toward that end, the investigators will evaluate the cost-effectiveness of the intervention from the perspective of the provider, payor, and society. These cost-effectiveness ratios will help decision makers generate informed decisions about appropriate and cost-effective treatment for high-risk patients with type 2 diabetes.
3. Study Population: Patients with Type 2 diabetes, older than 18 years of age, will be identified based on billing data (two visits with ICD-9 code of 250.xx in the preceding year) and subsequent chart review from nine Hershey Medical Center (HMC) primary care clinics and three Reading Hospital-affiliated primary care sites.
4. Major Inclusion Criteria: Inclusion criteria: Type 2 diabetes, age >18 who are at high risk based on any one of the following criteria: HbA1C >8.5, LDL >130, or BP >140/90.
5. Allocation to Groups: a stratified group randomization scheme whereby all patients being seen by the same doctor will be randomized to the same treatment group. The randomization will also be stratified by clinic site and size of doctor's practice. One group will be seen by nurse care managers, the other will continue with standard care.
6. Summary of Procedures: An initial pilot study will be performed with 60 patients from HMC and Reading Hospital clinics, for 2 months. This will consist of nurse case management intervention and feedback from the subjects to improve the study design. Subjects will be seen at 2, 4, 6 and 8 weeks. This study will end with focus groups of subjects to give their input as to what they did or did not like about the study, and how it might be improved. Pilot participants will have the option to enroll into the main study. No studies will be ordered for research purposes. Pregnancy screening will occur by verbally asking the subjects whether they believe they could be pregnant, since risk is very minimal.

   The main study will enroll 820 subjects at clinics from the Hershey Medical Center and Reading Hospital, with 2/3 of the subjects being enrolled at HMC, and 1/3 from the underserved Hispanic population. The study intervention will continue for 3 years. Patients will be enrolled into the nurse case management group or the control group dependent upon where they see their physician - randomization will occur in blocks based on clinics and physicians, not randomly per patient.

   In the main study, the intervention group patients will have an initial appointment with a nurse case manager (RN) (50 min) to review medical history, medications and control of diabetes and co-morbidities. A plan with patient specific treatment goals will be set up at this appointment. The patients will have follow up appointment set up for 2,4, and 6 weeks to review their progress, obtain standard diabetes laboratories and make necessary medication adjustments. The patients then will be seen by a nurse case manager on average once every 2-3 months, and a minimum of every 6 months, depending on their diabetes control. They will also continue to see their PCP (as scheduled per their PCP, normally once every 3-4 months). The control group patients will continue to follow with their PCP as scheduled, there will be no change from their usual care. The patients in both groups will be asked to complete 4 questionnaires (5 if they are depressed) assessing their emotional stress with diabetes, quality of life and treatment satisfaction at baseline and yearly for the study duration (3 years). Subjects will be randomly audio taped to ensure nurse case managers are following recommended guidelines of the research.

   Study outcomes such as HbA1c, lipids, blood pressure will be evaluated at baseline and then yearly in all patients. No laboratories will be done specifically for research purposes. The data will be extracted from the Penn State Diabetes Center Registry and charts (if required).

   For cost analysis, the investigators will be tracking outpatient and inpatient costs at the Hershey Medical Center and the Reading hospitals. In addition, the investigators will be tracking hospitalization costs outside of the hospitals by obtaining records from an existing registry managed by the State of Pennsylvania (the Pennsylvania Health Cost Containment Council), identified by social security numbers. This information along with all other information in the study will be safeguarded with strict confidentiality.
7. Major Risks & Discomforts: 1. Loss of confidentiality. 2. increased risk of low blood sugars with improved glycemic control, therefore the patients will be asked to test glucose on a regular basis - 2 -5 times daily, depending on their diabetes regimen. They will have a 24-hour contact phone number, specific to their primary care clinic, to call if problems arise.
8. Confidentiality: All research records, including those of subjects from Reading clinics, will be coded and kept at HMC. All consent forms will be forwarded to HMC. Records, audio tapes and the code key will be kept in the Endocrinology office in a locked file accessible only by the investigators.
9. Study Site Location(s): University Physician Health Groups (UPHG) is made up of 10 practice sites. For the purpose of this project 6 of the 10 HMC practice sites will participate and 3 of the Reading Hospital-affiliated ambulatory sites. All 3 sites are owned by The Reading Hospital and Medical Center, a non-profit hospital and health care organization.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* age > 18 years old who are at high risk based on any one of the following criteria:

  * HbA1C > 8.5
  * LDL > 130
  * BP > 140/90 within the last 6 months

Exclusion Criteria:

* patients who are pregnant upon entry in the study (however if a patient becomes pregnant in the course of the study, she can continue with the study)
* unable to communicate in either English or Spanish
* in nursing homes (and therefore unable to attend outpatient visits)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2006-08-10 (Actual); Primary Completion 2011-07-27 (Actual); Study Completion 2011-07-27 (Actual)

PRIMARY OUTCOMES:
% of patients reaching goal HbA1C (<7) | 2 years after enrollment
% of patients with BP goal (<130/80) | Two years after enrollment
% of patients with LDL at goal (<100) | 2 years after enrollment
% of patients at goal for all three parameters (HbA1C <7, BP <130/80, LDL <100) | 2 years after enrollment

SECONDARY OUTCOMES:
% of patients with yearly ophthalmologic exam | 2 years after enrollment
% of patients with yearly foot exam | 2 years after enrollment
% of patients with assessment for nephropathy | 2 years after enrollment
% of patients with nephropathy on ACE inhibitor or ARB | 2 years after enrollment
% of patients on aspirin | 2 years after enrollment
% of patients at or above CES-D depression score 16 for severe depression | 2 years after enrollment
Change in weight | 2 years after enrollment
Emotional distress (PAID survey) | 2 years after enrollment
Diabetes specific quality of life (ADD QOL) | 2 years after enrollment
Diabetes self care activities survey | 2 years after enrollment
Patient satisfaction survey (DTSQ) | 2 years after enrollment
Costs and cost-effectiveness | 2 years after enrollment
Physician satisfaction - survey filled out by physician | 2 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gabbay, MD, PhD, Principal Investigator — Penn State College of Medicine
Locations (2):
- United States (2):
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Reading Hospital, Reading, Pennsylvania

REFERENCES:
- [Background] Gabbay RA, Lendel I, Saleem TM, Shaeffer G, Adelman AM, Mauger DT, Collins M, Polomano RC. Nurse case management improves blood pressure, emotional distress and diabetes complication screening. Diabetes Res Clin Pract. 2006 Jan;71(1):28-35. doi: 10.1016/j.diabres.2005.05.002. Epub 2005 Jul 12. PMID 16019102
- [Derived] Stuckey HL, Dellasega C, Graber NJ, Mauger DT, Lendel I, Gabbay RA. Diabetes nurse case management and motivational interviewing for change (DYNAMIC): study design and baseline characteristics in the Chronic Care Model for type 2 diabetes. Contemp Clin Trials. 2009 Jul;30(4):366-74. doi: 10.1016/j.cct.2009.03.002. Epub 2009 Mar 26. PMID 19328244